Title: Product Testing of the FaceView Mask™: Usability Survey

PI: Samuel R. Atcherson, Ph.D.

**Study Title**: Product Testing of the FaceView Mask™: Usability Survey

**Principal Investigator**: Samuel R. Atcherson, Ph.D.

Department of Audiology and Speech Pathology

College of Health Professions

University of Arkansas for Medical Sciences

4301 W. Markham Street, Slot # 711

Little Rock, AR 72205
Telephone: 501.686.6860
Email: <a href="mailto:sratcherson@uams.edu">sratcherson@uams.edu</a>

**Study location**: University of Arkansas for Medical Sciences

4301 W. Markham Street Little Rock, AR 72205

## **Data Analysis**

As this is a product survey, and not a treatment or intervention project, all data will be reported using descriptive statistics in the aggregate.

Version #: 8.0 Date: 1.13.2023

Protocol template version dated 10.27.2020